CLINICAL TRIAL: NCT06189976
Title: Rapid Atrial Pacing After TAVI as a Predictor of Permanent Pacemaker Implantation
Brief Title: Rapid Atrial Pacing After TAVI to Predict Pacemaker Implantation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Leonidas Koliastasis, Interventional Cardiology Fellow, National and Kapodistrian University of Athens
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RAP-TAVI
Record Dates: First submitted 2023-12-17; First posted 2024-01-05 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Aortic Valve Disease; Transcatheter Aortic Valve Implantation; TAVI
Keywords: TAVR; TAVI; Rapid atrial pacing; Aortic stenosis
MeSH Terms: conditions — Aortic Valve Disease; Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rapid atrial pacing (Other): Diagnostic test group (single group)
  Interventions: Diagnostic Test: Rapid atrial pacing

INTERVENTIONS:
Diagnostic Test: Rapid atrial pacing — Rapid atrial pacing after TAVI

SUMMARY:
Despite Transcatheter aortic valve implantation (TAVI) evolution regarding techniques, equipment and experience, the need for permanent pacemaker implantation (PPI) post-TAVI remains an important drawback. The electrophysiology testing to stratify the risk or necessity of PPI post-TAVI is endorsed by the up-to-date guidelines and consensus documents and it is a valuable cut-off based method. Part of the answer is maybe hidden in the easy and applicable testing of the atrioventricular conduction system through rapid atrial pacing (RAP) with a common temporary pacemaker lead. This trial is designed to investigate the role and value of RAP after TAVI as a predictor of the necessity of new PPI.

DETAILED DESCRIPTION:
1. INTRODUCTION AND RATIONALE Despite Transcatheter aortic valve implantation (TAVI) evolution regarding techniques, equipment and experience, the need for permanent pacemaker implantation (PPI) post-TAVI remains an important drawback. PPI rates range widely from 7.8% to 20.3% based on the CENTER collaboration results, whereas significant differences are observed among the available devices. Except for hospitalization prolongation and higher costs, the impact of PPI in long term follow-ups seems to not to be innocent as it is associated with increased all-cause mortality and rehospitalization rates according to a recent meta-analysis. Data from the SWEEDHEART registry demonstrated no difference in survival in a median follow-up of 2.7 years, however as TAVI is offered to younger patients the long-term impact of PPI needs to be thoroughly investigated.

   The electrophysiology testing to stratify the risk or necessity of PPI post-TAVI is endorsed by the up-to-date guidelines and consensus documents and it is a valuable cut-off based method. Despite individualization is essential, thresholds provide added security and aid on final decisions. Variable HV intervals have been evaluated in clinical trials; 70ms is supported by ESC guidelines, while 55 in the presence of left bundle branch block in an observational trial. HV interval measurement seems appealing, but there is lack of cut-off consensus, not every Cath lab is equipped with electrophysiologic test equipment and TAVI operators are not generally familiar with these procedures.

   Part of the answer is maybe hidden in the easy and applicable testing of the atrioventricular conduction system through rapid atrial pacing (RAP) with a common temporary pacemaker lead. Krishnaswamy et al. performed post-TAVI atrial pacing from 70 to 120 beats/min in 284 patients and concluded that those who did not develop pacing-induced Wenckebach atrioventricular block exhibited very low probability of PPI. On the contrary, a recent report from Tan et al., found that atrial pacing-induced Wenckebach pre or post-TAVI in a total of 253 patients did not predict PPI. In this trial balloon expandable valves were used that are associated with lower rates of PPI and it is possible that larger sample size is needed for safe conclusions.
2. STUDY PROCEDURES TAVI will be planned to be performed with a temporary pacemaker lead in the right ventricle as a back-up for high grade conduction abnormalities or/and for on demand pacing. Before the procedure initiation, if the patient is stable and not pacemaker-dependant the temporary pacemaker electrode will be placed into the right atrium. This manoeuvre adds no cost and no additional risk for the patient as the electrode is already placed in the right chambers. Surface electrocardiogram will be recorded at the whole procedure. Atrial pacing will be initiated till Wenckebach AV block is observed and recorded or till the maximum atrial pacing rate is reached. The rate that AV block was observed will be catalogued. Maximum atrial pacing rate will be 150 beats/min (cycle length 400ms). After a successful TAVI procedure, if the patient is stable and not pacemaker-dependant the temporary pacemaker electrode will be placed again into the right atrium. The RAP test will be performed again.
3. STUDY MONITORING 3.1 Responsibility of the investigators The investigators undertake to perform the study in accordance with this protocol and GCP. For the trial duration, the investigator(s) will maintain complete and accurate documentation including - but not limited to - medical records, trial progress records, laboratory reports, case report forms, signed informed consent forms, device accountability records, correspondence with the IRB, adverse event reports, and information regarding patient discontinuation or completion of the trial.

   3.2 Case report forms It is the responsibility of the investigator to maintain an accurate CRF to record all observations and other data pertinent to the clinical and laboratory investigations. All CRF should be completed in their entirety in a neat, legible manner to ensure accurate interpretation of data. The data may be recorded either on hard copies or electronic data capture. This data will be monitored by and forwarded to the primary investigator (PI) in an expedited fashion.
4. ADVERSE EVENTS All events will be registered in the CRF as defined by GCP. Adverse events will be actively checked during follow-up. Patient folder will provide contact information for patients in case of questions and when complications occur. Any complication will be managed at each centre per local practice.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥18 years old.
2. Patient understands the purpose, the potential risks as well as benefits of the trial and is willing to participate in all parts of the follow-up.
3. Patient has given written consent to participate in the trial.
4. Patients undergoing TAVI as a treatment of severe aortic stenosis (AS).
5. Patient in sinus rhythm.
6. Patients planned for TAVI with utilization of temporary pacemaker electrode placement.

Exclusion Criteria:

1. Ongoing infection, including active endocarditis.
2. Implanted permanent pacemaker and/or implantable cardioverter/defibrillator.
3. Patients developing persistent second or third degree atrioventricular block (AV) after TAVI.
4. Underlying rhythm other than sinus based on the surface ECG leads monitoring after TAVI.
5. Patients with second or third degree AV block identifyied on the screening pre-TAVI ECG.
6. Enrolment in another study that competes or interferes with this study.
7. Subject will not be able to comply with the follow-up requirements according to investigators' opinion.
8. Pregnant or breast-feeding females or females who intend to become pregnant during the time of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Permanent pacemaker implantation rates | 30 days
  Rates of permanent pacemaker implantation after TAVI

SECONDARY OUTCOMES:
Mortality rates | 30 days
  Rates of mortality after TAVI
Mortality rates | 6 months
  Rates of mortality after TAVI
Permanent pacemaker implantation rates | 6 months
  Rates of permanent pacemaker implantation after TAVI
Mortality rates | 12 months
  Rates of mortality after TAVI
Permanent pacemaker implantation rates | 12 months
  Rates of permanent pacemaker implantation after TAVI

CONTACTS AND LOCATIONS:
Overall Officials: Leonidas Koliastasis, Principal Investigator — National and Kapodistrian University of Athens
Locations (2):
- CHU Saint-Pierre, Brussels, Belgium
- Hippocration Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Knecht S, Schaer B, Reichlin T, Spies F, Madaffari A, Vischer A, Fahrni G, Jeger R, Kaiser C, Osswald S, Sticherling C, Kuhne M. Electrophysiology Testing to Stratify Patients With Left Bundle Branch Block After Transcatheter Aortic Valve Implantation. J Am Heart Assoc. 2020 Mar 3;9(5):e014446. doi: 10.1161/JAHA.119.014446. Epub 2020 Feb 22. PMID 32089049
- [Result] Krishnaswamy A, Sammour Y, Mangieri A, Kadri A, Karrthik A, Banerjee K, Kaur M, Giannini F, Pagliaro B, Ancona M, Pagnesi M, Laricchia A, Weisz G, Lyden M, Bazarbashi N, Gad M, Ahuja K, Mick S, Svensson L, Puri R, Reed G, Rickard J, Colombo A, Kapadia S, Latib A. The Utility of Rapid Atrial Pacing Immediately Post-TAVR to Predict the Need for Pacemaker Implantation. JACC Cardiovasc Interv. 2020 May 11;13(9):1046-1054. doi: 10.1016/j.jcin.2020.01.215. Epub 2020 Apr 15. PMID 32305392
- [Result] Tan BE, Hashem A, Boppana LKT, Mohamed MS, Abbas SF, Faisaluddin M, Thakkar S, Ahmed AK, Hall C, Abtahian F, Rao M, Bhatt DL, Depta JP. Utility of rapid atrial pacing before and after TAVR with balloon-expandable valve in predicting permanent pacemaker implantation. Catheter Cardiovasc Interv. 2023 Nov;102(5):919-928. doi: 10.1002/ccd.30817. Epub 2023 Sep 12. PMID 37698294
- [Derived] Koliastasis L, Doundoulakis I, Tsiachris D, Pannone L, Skalidis I, de Hemptinne Q, Xaplanteris P, Toutouzas K, de Asmundis C. Rapid Atrial Pacing After TAVI for Pacemaker Prediction. Rev Cardiovasc Med. 2025 Aug 15;26(8):39074. doi: 10.31083/RCM39074. eCollection 2025 Aug. PMID 40927105